CLINICAL TRIAL: NCT00452075
Title: A Phase II Study of Erlotinib and Predictive Markers as First-line Treatment of Advanced Non-small Cell Lung Cancer for Patients Unfit for Chemotherapy
Brief Title: Erlotinib as First-line Treatment of Advanced Non-small Cell Lung Cancer (NSCLC) for Patients Unfit for Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Gedske Daugaard, Professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 20539
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR expression; erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm 1 medicine (Experimental): erlotinib daily
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — 150mg daily
  Other Names: tarceva

SUMMARY:
A phase II study of Tarceva (Erlotinib) and predictive markers as first-line treatment of advanced non-small cell lung cancer for patients unfit for chemotherapy (NSCLC) Clinical Phase II Stage IIIB or IV non-small cell lung cancer (NSCLC) Primary end point: Disease control rate (= CR+PR and SD at 8 weeks /patients). Secondary end point: Safety (Serious Adverse Events, Adverse Events leading to premature withdrawal, unexpected TarcevaTM related AEs) .Correlation of EGFR expression rate (HER1) and FISH potentially predictive for response.

An open-label, non randomized, multicenter, clinical trial of TarcevaTM as single agent The sample size is 29 patients in 2 stages and based on Simon´s optimal 2 stage design. Stage 1 will accrue 10 patients, if less than 1 response is observed the study will stop; if more than 1 response is observed the accrual will continue up till 29 patients. A total of 29 patients would be entered and the treatment will be declared to have sufficient activity to deserve further attention if at least 5 patients obtain disease control.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented diagnosis of inoperable, locally advanced, recurrent or metastatic (Stage IIIB or Stage IV) NSCLC.
* Chemo-naïve patients.
* Patients who are in the investigator's opinion not medically suitable for chemotherapy.
* Measurable disease according to the RECIST criteria.
* ECOG performance status of 0 - 3.
* Life expectancy of at least 12 weeks.
* Patients must be able to take oral medication.
* Serum calcium within normal ranges
* ≥ 4 weeks since prior surgery or radiation therapy
* For all females of childbearing potential a negative pregnancy test must be obtained within 48 hours before starting therapy and must use effective contraception
* 18 years of age or older
* Written (signed) Informed Consent to participate in the study

Exclusion Criteria:

* Prior systemic antitumor therapy
* Any unstable systemic disease which according to the investigator contraindicates the use of the study drug render the subject at high risk from treatment complications (including active infection, unstable angina, myocardial infarction within the previous month, inflammatory bowel disease, hepatic disease with serum bilirubin ≥ 2 upper limit of normal (ULN) or AST and/or ALT ≥ 2 x ULN (or ≥ 5 x ULN if clearly attributable to liver metastasis), renal disease with acute renal failure or serum creatinine ≥ 5 x ULN.
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Nursing mothers or pregnant woman.
* Hypersensitivity to Tarceva or co-formulants.
* Patients with brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation.
* Patients with brain metastasis or spinal cord compression that not are in a stable condition despite treatment with steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 2010

SECONDARY OUTCOMES:
To investigate the tolerability and safety of erlotinib in patients, who can not receive chemotherapy, by registration of side-effects. | 2010
Correlation of EGFR expression rate and FISH potentially predictive for response | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Pappot Helle, MD, DMSC, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Department of Oncology, Århus University Hospital, Aarhus
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Department of Oncology, Odense University Hospital, Odense